CLINICAL TRIAL: NCT04709874
Title: Paravertebral Block Versus Suprascapular Block for Treatment of Frozen Shoulder: a Prospective, Randomized Clinical Trial
Brief Title: Paravertebral Block vs. Suprascapular Block for Treatment of Frozen Shoulder
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Zoher Naja, Anesthiologist, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11012021
Record Dates: First submitted 2021-01-12; First posted 2021-01-14 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Pain, Shoulder
MeSH Terms: conditions — Shoulder Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Paravertebral block (Experimental): Patients will receive paravertebral block guided by a nerve stimulator.
  Interventions: Other: Paravertebral block
- Suprascapular block (Active Comparator): Patients will receive suprascapular block
  Interventions: Other: Suprascapular block

INTERVENTIONS:
Other: Paravertebral block — Paravertebral block using nerve stimulator guidance will be done at C7-T1
  Arms: Paravertebral block
Other: Suprascapular block — Paravertebral block using nerve stimulator guidance will be done
  Arms: Suprascapular block

SUMMARY:
Background: Adhesive capsulitis, or frozen shoulder, is a major orthopedic condition that causes pain and functional limitation. Although different nonsurgical conservative therapies such as physical therapy, nonsteroidal anti-inflammatory drugs, and corticosteroid injections have been used, yet there is no standard treatment for frozen shoulder.

Objectives: The primary objective of this study is to compare the effectiveness of nerve stimulator guided paravertebral block versus suprascapular block for treatment of frozen shoulder. The primary outcome is pain measured through the Visual Analogue Scale (VAS) over a follow up period of 6 months.

Methods: This is a prospective randomized clinical trial that will be conducted between February 2021 and January 2022. Patients will be randomly allocated into two groups. Group I will receive paravertebral block guided by a nerve stimulator. Group II patients will receive suprascapular nerve block. Patients will be followed up at week 1, month 1, month 3 and month 6.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* presenting with frozen shoulder and were unresponsive to conservative therapy

Exclusion Criteria:

* Complete rotator cuff tear
* Osteoarthritis
* Calcified tendinitis
* History of shoulder joint injury
* Cervical radiculopathy
* Bleeding disorder
* Active infection
* Allergy to Bupivacaine
* Diabetes Mellitus

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-02 (Actual); Primary Completion 2023-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
Pain score | 6 months
  Pain will measured through the Visual Analogue Scale (VAS). 0 indicates no pain and 10 indicates maximum pain

CONTACTS AND LOCATIONS:
Overall Officials: Zoher Naja, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon